CLINICAL TRIAL: NCT06276153
Title: Construction of Multicenter Retrospective Registry Cohort Database for Gallbladder Cancer
Acronym: CRGGCext
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liu Ying-bin, Director of Pancreato-biliary Surgery, Principal Investigator, Professor, RenJi Hospital
Other Study IDs: CRGGCext
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Biliary Tract Diseases; Gallbladder Cancer; Gallbladder Neoplasms
Keywords: gallbladder cancer; gallbladder neoplasms; cohort study; registry cohort; biliary tract neoplasms
MeSH Terms: conditions — Biliary Tract Diseases; Gallbladder Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gallbladder cancer: Diagnostic criteria:
  Patients with gallbladder cancer diagnosed by pathology, and combined with clinical manifestations and imaging results, the first diagnosis and discharge were diagnosed as patients with gallbladder cancer.
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — retrospective registry cohort with no other specific interventions

SUMMARY:
The aim of the study is to establishing a standardized clinical information database for patients with malignant tumors of gallbaldder. Based on the database, real-world clinical research on the diagnosis and treatment of biliary tract tumors is about to be carried out, and a high-standard cohort research foundation is laid for precision therapy.

DETAILED DESCRIPTION:
From the date of commencement of the study, patients who presented to the participating medical institutions in the study and were clinically diagnosed as gallbladder cancer, and who met the inclusion criteria and did not meet any of the exclusion criteria, were enrolled in the study cohort after signing an informed consent form.

The research objectives of this study mainly include establishing a structured dataset standard for gallbladder cancer based on the diagnosis and treatment norms and clinical pathways and carrying out clinical registration research on gallbladder cancer and build a specific disease cohort

The outcome indicators of this study included overall survival time OS, recurrence-free survival time PFS, R0 resection rate of patients treated with biliary malignancy, and objective response rate ORR. The main measurement indicators of this study include the patient's demographic information, past history, life history, admission, preoperative examination information, surgery, postoperative situation, discharge, follow-up, outcome indicators, routine examination results of biological samples and multi-omics sequencing results, the above data are derived from the original records of prospective case questionnaires, the original records of patients' electronic medical records and the examination results of patients' biological samples. The outcome of follow-up was defined as patients having been followed up for five years, or having a patient lost to follow-up or dying during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent, have good compliance, and be willing to accept follow-up and provide blood samples
* Age 18-74 years old, gender is not limited
* Clinical diagnosis of gallbladder cancer, including unoperated patients preliminarily diagnosed as gallbladder cancer according to the results of imaging examinations and laboratory tests, or pathological examination of patients treated with surgery confirmed as malignant tumors of the gallbladder.
* The primary tumor is located in gallbladder floor, gallbladder body, gallbladder neck or gallbladder duct.
* Karnofsky performance score greater than 50.

Exclusion Criteria:

* Patients with gallbladder cancer, gallbladder cancer foci are not primary lesions.
* Patients with gallbladder cancer, combined with serious central nervous system diseases, respiratory diseases, autoimmune diseases, chronic renal insufficiency and other diseases, long-term use of immunosuppressants, combined with serious uncontrolled infections.
* Patients with gallbladder cancer, who also have active cardiovascular and cerebrovascular diseases, have cerebrovascular accidents, myocardial infarction, unstable angina pectoris, or grade II. or above congestive heart failure according to the standards of the New York Heart Association, and require serious arrhythmias requiring drug treatment.
* Patients with gallbladder cancer, women of childbearing age who have a positive blood pregnancy test or have not had a pregnancy test, pregnant or breastfeeding women.
* The patient is participating in other therapeutic clinical trials where treatment measures cannot be clarified or treatment information cannot be collected .

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gallbladder cancer diagnosed by pathology, and combined with clinical manifestations and imaging results, the first diagnosis and discharge were diagnosed as patients with gallbladder cancer.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of enrollment until the date of death from any cause, whichever came first, assessed up to 5-years.
  OS in patients with biliary malignancies was long-term follow-up data, defined as the primary endpoint, OS is calculated from the date of surgery for patients treated surgically, and OS is calculated from the date of diagnosis for patients treated non-surgically. The expected survival of patients with benign biliary tumors is longer, and this study does not select the study endpoint based on the follow-up of patients with benign biliary tumors, but mainly collects perioperative diagnosis and treatment data and collects biological samples.

SECONDARY OUTCOMES:
progression-free survival | From date of enrollment until the date of first documented progression from any cause, whichever came first, assessed up to 5-years.
  PFS was defined as a secondary endpoint. PFS is calculated from the date of surgery for patients treated surgically, and PFS is calculated from the date of diagnosis for patients treated non-surgically. The expected survival of patients with benign biliary tumors is longer, and this study does not select the study endpoint based on the follow-up of patients with benign biliary tumors, but mainly collects perioperative diagnosis and treatment data and collects biological samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Bin Liu, PhD., Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No